CLINICAL TRIAL: NCT02560857
Title: Clinical Evaluation of Quantiferon-Monitor to Predict Outcomes in Solid Organ Transplant Recipients
Acronym: QTF-Monitor
Status: Completed | Type: Observational
Sponsor: Deepali Kumar (Other)
Responsible Party: Sponsor-Investigator, Deepali Kumar, Physician, Transplant Infectious Diseases, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 14-8133
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Immunity, Cellular
Keywords: Quantiferon-Monitor; organ rejection; global immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples (plasma will be extracted to perform Quantiferon-Monitor test)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Quantiferon-Monitor assay — The QFT-Monitor assay is a recently developed non-pathogen specific immune assay based on immune activation of both innate and adaptive immunity.

SUMMARY:
The study will prospectively determine the clinical utility of non-pathogen specific cellular immunity assessment using the Quantiferon-Monitor to quantify the degree of immunosuppression. The investigators will use the results of the assay to predict whether patients develop opportunistic infections and predict organ rejection.

DETAILED DESCRIPTION:
Solid organ transplant (SOT) recipients undergo life-long immunosuppression to prevent allograft rejection. However, this also puts patients at significant risk for opportunistic infection. The degree of immunosuppression varies for each individual and is likely influenced by a combination of clinical factors such as antirejection medication, comorbidities, patient age as well as the state of patient immune system. Thus far, there have been no standardized methods to quantify the degree of global immunosuppression. A new blood test (Quantiferon-Monitor) has been recently developed that might help predict the level of immune suppression. The purpose of this study is to determine whether this new test will help determine a person's level of immune suppression after organ transplant. This will be done by trying to relate the level of immunity with the development of infection or rejection. If the test for immunosuppression is helpful, it may help us to better take into account the differences in patients when designing therapy. Ultimately, it may help develop better ways for preventing infections and transplant rejections.

ELIGIBILITY:
Inclusion Criteria:

* Adult SOT recipients on at least one immunosuppressive medication able to comply with the protocol.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult SOT recipients on at least one immunosuppressive medication.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of participants that develop Opportunistic infections | 1 year
  The results of the assay will be used to predict whether patients develop opportunistic infections.

SECONDARY OUTCOMES:
Number of participants that develop Acute cellular rejection | 1 year
  The results of the assay will be used to predict whether patients develop acute cellular rejection.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada